CLINICAL TRIAL: NCT02408146
Title: The Effect of Parecoxib Sodium Intravenous Patient-controlled Analgesia in Laparotomic Liver Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lianxin-001
Record Dates: First submitted 2014-04-01; First posted 2015-04-03 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2014-03

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — parecoxib; Saline Solution; Celecoxib

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (3):
- conventional intravenous infusion pump (Experimental): The first group receives conventional intravenous infusion pump of patient-controlled analgesia.
  Interventions: Procedure: conventional intravenous infusion pump; Drug: fentanyl citrate+ ondansetron hydrochloride + normal saline
- parecoxib (Experimental): The second group has oral celecoxib before surgery, then receives parecoxib sodium intravenously guttae after surgery.
  Interventions: Drug: parecoxib; Drug: celecoxib
- new intravenous infusion pump (Experimental): The third group uses new intravenous infusion pump of patient-controlled analgesia after surgery.
  Interventions: Drug: parecoxib; Procedure: intravenous infusion pump of patient-controlled analgesia; Drug: celecoxib

INTERVENTIONS:
Procedure: conventional intravenous infusion pump — The first group receives conventional intravenous infusion pump of patient-controlled analgesia (fentanyl citrate 20 mg/mL/kg + ondansetron hydrochloride 16 mg/8 mL + normal saline) for three days after surgery. The pump is infused continuously at the basic flow rate of 2 mL/h, 0.5 mL of bolus can be injected if the patients press the button once upon experiencing pain. The lock-out time for each bolus injection is 15 minutes.
  Arms: conventional intravenous infusion pump
Drug: parecoxib — The second group has oral celecoxib before surgery, then receives 40 mg parecoxib sodium intravenously guttae twice a day for three days after surgery.
  Other Names: CAS number: 202409-33-4
  Arms: new intravenous infusion pump; parecoxib
Procedure: intravenous infusion pump of patient-controlled analgesia — The third group has oral celecoxib before surgery, and receives 40 mg parecoxib sodium intravenously guttae immediately after surgery, then uses new intravenous infusion pump of patient-controlled analgesia (parecoxib sodium 1 mg/mL + normal saline) for three days after surgery. The pump is infused continuously at the basic flow rate of 2 mL/h, 0.5 mL of bolus can be injected if the patients press the button once upon experiencing pain. The lock-out time for each bolus injection is 15 minutes.
  Arms: new intravenous infusion pump
Drug: fentanyl citrate+ ondansetron hydrochloride + normal saline
  Arms: conventional intravenous infusion pump
Drug: celecoxib
  Arms: new intravenous infusion pump; parecoxib

SUMMARY:
The investigators hypothesized that using new intravenous infusion pump of patient-controlled analgesia (parecoxib sodium 1 mg/mL + normal saline) would significantly improve postoperative pain control compare to conventional intravenous infusion pump of patient-controlled analgesia (fentanyl citrate 20 mg/mL/kg + ondansetron hydrochloride 16 mg/8 mL + normal saline). This prospective randomized controlled trial was designed to evaluate the benefit of new intravenous infusion pump of patient-controlled analgesia (parecoxib sodium 1 mg/mL + normal saline) for postoperative analgesia after laparotomic liver resection.

ELIGIBILITY:
Inclusion Criteria:

Patients need laparotomic liver resection.

Exclusion Criteria:

Patients with contraindications to spinal anesthesia or intrathecal morphine, difficulty understanding passive cutaneous anaphylaxis, a history of drug dependence or chronic pain, body mass index greater than 35 kg/m2, or history of sleep apnea were excluded from this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
The measure is a composite outcome measure consisting of multiple measures,pain scores, sedation, nausea, pruritus, and respiratory rate. | With or without changes in the three days after surgery
  Pain scores are evaluated with a visual analog scale of 0 to 100 and are measured at rest and with movement such as cough or incentive spirometry at 6, 9, 12, 18, 24, 36, 48 and 72 hours. Sedation, nausea, and pruritus are also measured at 6, 9, 12, 18, 24, 36, 48 and 72 hours. All the measures count together to get a composite outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- harbin Medical University, Harbin, Heilongjiang, China